CLINICAL TRIAL: NCT01153373
Title: The Dynamic Assessment and Referral System for Substance Abuse: Evaluation
Brief Title: Dynamic Assessment and Referral System - Evaluation
Acronym: DARSSA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Edwin Boudreaux, Study Principle Investigator, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: H-13419
Record Dates: First submitted 2010-06-24; First posted 2010-06-30 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Smoking; Alcohol Abuse; Drug Abuse
Keywords: Detection of tobacco, alcohol, and drug use.
MeSH Terms: conditions — Smoking; Alcoholism; Substance-Related Disorders | interventions — Tobacco Products; Ethanol; Counseling

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Minimal Intervention Control (Placebo Comparator): All patients that give consent to participate in the study ("participants") who are randomly assigned to the control condition will complete the computerized DARSSA for assessment purposes only. The reports will not be printed or dynamic referrals generated, and all patients will receive treatment-as-usual by their ED providers.
  Interventions: Behavioral: Self-administered computerized assessment for tobacco, substance abuse, and alcohol use.
- DARSSA Intervention (Active Comparator): All participants randomized to the DARSSA Intervention will be given instructions for how to complete the assessment. Once completed, the treating emergency physician will be expected to (1) give substance using patients the Patient Feedback Report, (2) recommend they review it carefully, and (3) encourage them to consider following up with the referrals.
  Interventions: Behavioral: Self-Administered Computerized Assessment and Counseling for Tobacco, Alcohol, and Substance Abuse

INTERVENTIONS:
Behavioral: Self-administered computerized assessment for tobacco, substance abuse, and alcohol use. — All patients that give consent to participate in the study ("participants") who are randomly assigned to the control condition will complete the computerized DARSSA for assessment purposes only.
  Arms: Minimal Intervention Control
Behavioral: Self-Administered Computerized Assessment and Counseling for Tobacco, Alcohol, and Substance Abuse — All participants randomized to the DARSSA Intervention will be given instructions for how to complete the assessment. Once completed, the treating emergency physician will be expected to (1) give substance using patients the Patient Feedback Report, (2) recommend they review it carefully, and (3) encourage them to consider following up with the referrals.
  Arms: DARSSA Intervention

SUMMARY:
The investigators study will use a randomized controlled design. Eligible and consenting participants will be randomly assigned to one of two conditions: (1) DARSSA Intervention condition, or (2) Minimal Intervention Control condition. All enrolled participants will undergo the DARSSA baseline assessment and will be interviewed immediately following their ED discharge to assess relevant outcomes, such as whether they were asked about substance use and given a referral during their visit. This is referred to as the post-visit interview. All risky substance users enrolled during all phases will be interviewed again at 1- and 3-months post-visit to assess substance use, treatment engagement, and other outcomes. The primary difference between the two conditions is that, for the DARSSA Intervention condition, the subjects will have their reports printed and will be given the option of receiving the dynamic referral, while for the Minimal Intervention Control condition the subjects will undergo the assessment and will receive the standard substance abuse treatment referral list currently in use clinically at each site. The number of assessments and interactions with research staff will remain equal between the two conditions, with the only difference being the active intervention of the DARSSA reports and referrals, and any counseling by healthcare providers this engenders. The remainder of this section describes each phase of the study and enrollment procedures.

DETAILED DESCRIPTION:
Screening process. All patients who verbally consent to being screened by the RA will undergo a computer assisted screening for substance abuse (Rapid Screener) administered by the research assistant. Patients who use tobacco, misuse alcohol, or use illicit drugs will be further screened for eligibility to participate in the randomized trial. Eligible patients will be invited to participate and will sign the consent form. Participants will then be assigned to one of the two conditions by the computer using a random number generator. Results obtained as part of the Rapid Screener will be for research purposes only. They will not be reported to healthcare providers, unless the participant is enrolled into the study and is assigned to the DARSSA Intervention condition (see below).

Minimal Intervention Control. All patients that give consent to participate in the study ("participants") who are randomly assigned to the control condition will complete the computerized DARSSA for assessment purposes only. The reports will not be printed or dynamic referrals generated, and all patients will receive treatment-as-usual by their ED providers. This will preserve the treatment-as-usual nature of the baseline while maintaining consistency in the administration of the DARSSA between phases of the study. Although ED clinicians will know that a study is being conducted in the ED, they will not be informed of the results of the research assessment, nor will they be given any instruction or training beforehand to change their standard screening, counseling, and referral practices. This means that substance use screening is likely to be inconsistent and counseling or referrals by provider rare. To maintain ethical standards, the RAs will provide a substance abuse treatment resource list (passive referral list) to all subjects who screen positive, even though this often does not happen during routine clinical practice. Additionally, suicidal ideation is not directly assessed as part of the study, but it is possible that participants will spontaneously report suicidal ideation. If this happens, the RA will notify the treating physician. Both of these efforts could conceivably introduce interventions the patient may not otherwise have received, but there is no viable alternative if the investigators are to ensure patient safety.

DARSSA Intervention. All participants randomized to the DARSSA Intervention will be given instructions for how to complete the assessment. Since the DARSSA is self-administered and, like all Polaris products, does not require computer literacy, instructions will be simple and do not require a clinician to administer. Once completed, the treating emergency physician will be expected to (1) give substance using patients the Patient Feedback Report, (2) recommend they review it carefully, and (3) encourage them to consider following up with the referrals. Any additional assessment or counseling will be optional and left to individual provider practice. We considered creating a standardized counseling protocol but decided against it. We want to maintain an ecologically valid evaluation. In the "real world," providers would not be given extensive health behavior counseling training or asked to follow a standardized counseling protocol when implementing the DARSSA. Training providers on health behavior counseling would act as an additional intervention in its own right, and it could potentially mask our ability to determine what effect the DARSSA alone is having.

ELIGIBILITY:
Inclusion Criteria:

- Age 18 years or older and receiving treatment in the ED

Exclusion Criteria:

* sustained altered mental status (e.g., psychosis, delirium, disorientation, unresponsive)
* hostile or agitated behavior
* sexual assault victims
* trauma patients who are on backboards or who must remain supine
* severe illness that would preclude conversation or interface with a computer (e.g., intubation, persistent vomiting, severe pain)
* or factors precluding follow-up, like transient residence or lack of a telephone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 758 (Actual)
Dates: Start 2010-06; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Prevalence of detected tobacco, alcohol, and drug use in emergency room patients. | November 2009 - June 2013
  When comparing the intervention (DARSSA) group to the treatment as usual group, is there an increase in the detected prevalence of tobacco use, alcohol use, and drug abuse.

SECONDARY OUTCOMES:
Increase in delivery of health care (i.e. - education/counseling/referral) for emergency room patients that report tobacco use, alcohol use, and/or substance abuse. | November 2009 - June 2013
  When the intervention (DARSSA) group is compared to the treatment as usual group, is there an increase in the amount of education/counseling/referral for emergency room patients who report tobacco use, alcohol use, and/or substance abuse.

CONTACTS AND LOCATIONS:
Overall Officials: Edwin Boudreaux, PhD, Principal Investigator — UMass Medical School
Locations (1):
- UMass Memorial Medical Center - university campus, Worcester, Massachusetts, United States

REFERENCES:
- [Derived] Haskins BL, Davis-Martin R, Abar B, Baumann BM, Harralson T, Boudreaux ED. Health Evaluation and Referral Assistant: A Randomized Controlled Trial of a Web-Based Screening, Brief Intervention, and Referral to Treatment System to Reduce Risky Alcohol Use Among Emergency Department Patients. J Med Internet Res. 2017 May 1;19(5):e119. doi: 10.2196/jmir.6812. PMID 28461283
- [Derived] Boudreaux ED, Abar B, Haskins B, Bauman B, Grissom G. Health evaluation and referral assistant: a randomized controlled trial to improve smoking cessation among emergency department patients. Addict Sci Clin Pract. 2015 Nov 5;10:24. doi: 10.1186/s13722-015-0045-2. PMID 26542471